CLINICAL TRIAL: NCT03028519
Title: Vitamin D, Leptin, Vitamin D Receptor Polymorphism, and Treatment-Related Morbidity in Ovarian Cancer
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Oklahoma (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 7488
Record Dates: First submitted 2017-01-10; First posted 2017-01-23 (Estimated); Last update posted 2022-04-19 (Actual); Status verified 2022-04

CONDITIONS: Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Cholecalciferol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (Experimental): Vitamin D levels will be measured at the time of routine blood work. If Vitamin D levels are found to be low, patients will take 50,000 IU of vitamin D3 weekly daily as maintenance therapy. There is no prospective control arm.
  Interventions: Drug: Vitamin D3

INTERVENTIONS:
Drug: Vitamin D3 — Vitamin D3

SUMMARY:
This study will evaluate serum vitamin D (25(OH)D) and serum leptin levels at the time of diagnosis of ovarian, primary peritoneal, and/or fallopian tube cancer as well as vitamin D receptor mutation status (FokI SNP genotype). The study will evaluate the impact of vitamin D repletion on serum vitamin D levels, serum leptin levels, and treatment-related morbidity in these patients.

DETAILED DESCRIPTION:
This study will contain 2 cohorts: those with normal serum 25(OH)D and those with low serum 25(OH)D at enrollment. The study will take place in women with ovarian, primary peritoneal, and fallopian tube cancer.

Patients who have given written consent to enroll in the study will have a serum 25(OH)D levels, serum leptin levels, and vitamin D receptor FokI single nucleotide polymorphism analyzed at the time of diagnosis. Patients with vitamin D deficiency will be prescribed vitamin D supplementation according to current guidelines. Treatment with cholecalciferol will not impact cancer therapy. Participants treatment course information will be collected prospectively, but will not be dictated by this study. Serum 25(OH)D and leptin levels will be collected again at the completion of primary therapy, 6 months after the completion of primary therapy, and at the time of disease recurrence. If patients remain vitamin D deficient at any of these follow-up time points, they will be referred to an endocrinologist for further work-up and treatment of their vitamin D deficiency. Data collection will continue for up to 1 year after enrollment.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a histologic diagnosis of ovarian, fallopian tube, or primary peritoneal carcinoma per pre-treatment biopsies by laparoscopy, or interventional radiology, paracentesis, or CT guided core biopsy. Histologic documentation of the original primary tumor is required via the pathology report.
* Patients must have adequate: Renal function: Glomerular Filtration Rate (GFR) > 30; Gastrointestinal absorption: No underlying malabsorption syndrome (i.e. inflammatory bowel disease, celiac disease)
* Ability to tolerate oral medication
* Patients taking vitamin D at the time of enrollment without a diagnosis of vitamin D deficiency
* Patients of childbearing potential must have a negative pregnancy test prior to the study entry and be practicing an effective form of contraception.
* If applicable, patients must discontinue breastfeeding prior to study entry.
* Patients must be at least 18 years old

Exclusion Criteria:

* Patients with a known pre-existing diagnosis of vitamin D deficiency.
* Patients with renal disease and a GFR <30
* Patients with primary hyperparathyroidism
* Patients with other invasive malignancies, with the exception of nonmelanoma skin cancer.
* Patients with concomitant endometrial cancer diagnosed at the time of their ovarian cancer are allowed to participate if the endometrial cancer is International Federation of Gynecology and Obstetrics stage 1B or less.
* Patients of childbearing potential, not practicing adequate contraception, patients who are pregnant, or patients who are breastfeeding are not eligible for this trial.

Ages: 18 Years to 99 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2017-01-31 (Actual); Primary Completion 2020-12-30 (Actual); Study Completion 2020-12-30 (Actual)

PRIMARY OUTCOMES:
Treatment Related Morbidity | 1 year
  Chemotherapy and 30-day post-operative surgical morbidity will be measured and reported in aggregate as number of patients with chemotherapy-related and/or surgery-related morbidity.

SECONDARY OUTCOMES:
Survival | 1 year
  disease free survival
Identify serum 25(OH)D and serum leptin relationship | baseline, at completion of primary cancer therapy, at 6 months post-completion of primary therapy, at recurrence or at 1 year post-completion of primary therapy
  Change in serum 25(OH)D levels with vitamin D repletion
Evaluate serum level changes | baseline, at completion of primary therapy, at 6 months post-completion of primary therapy, at recurrence or at 1 year post-completion of primary therapy]
  Change in serum Leptin levels with vitamin D repletion
Mutation Status | at time of enrollment
  Vitamin D Receptor FokI Single Nucleotide Polymorphism mutation status

CONTACTS AND LOCATIONS:
Overall Officials: Laura Holman, MD, Principal Investigator — University of Oklahoma
Locations (1):
- University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol (2021-09-09): https://cdn.clinicaltrials.gov/large-docs/19/NCT03028519/Prot_000.pdf
  • Statistical Analysis Plan (2021-07-01): https://cdn.clinicaltrials.gov/large-docs/19/NCT03028519/SAP_001.pdf